CLINICAL TRIAL: NCT05800015
Title: A Randomized, Double-Blind Phase 2/3 Study of Fianlimab (Anti-LAG-3 Antibody), Cemiplimab (Anti-PD-1 Antibody), and Chemotherapy Versus Cemiplimab and Chemotherapy in First-Line Treatment of Patients With Advanced Non-Small Cell Lung Cancer (NSCLC) Irrespective of PD-L1 Expression Levels
Brief Title: A Trial to Learn How the Combination of Fianlimab With Cemiplimab and Chemotherapy Works Compared With Cemiplimab and Chemotherapy for Treating Adult Patients With Advanced Non-small Cell Lung Cancer
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R3767-ONC-2236; 2022-501577-40-00 (EU CTIS Number)
Record Dates: First submitted 2023-03-23; First posted 2023-04-05 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Non-small Cell Lung Cancer
Keywords: NSCLC; Lung cancer; Programmed cell death ligand-1; PD-L1; Lymphocyte-activation gene 3; LAG-3; African descent
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — cemiplimab; Pemetrexed; Paclitaxel; Carboplatin; Cisplatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Phase 2 - Arm A (Experimental): Randomized 1:1:1 fianlimab (higher dose) + cemiplimab + platinum-doublet chemotherapy
  Interventions: Drug: fianlimab; Drug: cemiplimab; Drug: Pemetrexed; Drug: Paclitaxel; Drug: Carboplatin; Drug: Cisplatin
- Phase 2 - Arm B (Experimental): Randomized 1:1:1 fianlimab (lower dose) + cemiplimab + platinum-doublet chemotherapy
  Interventions: Drug: fianlimab; Drug: cemiplimab; Drug: Pemetrexed; Drug: Paclitaxel; Drug: Carboplatin; Drug: Cisplatin
- Phase 2 - Arm C (Experimental): Randomized 1:1:1 cemiplimab + platinum-doublet chemotherapy + placebo
  Interventions: Drug: cemiplimab; Drug: Pemetrexed; Drug: Paclitaxel; Drug: Carboplatin; Drug: Cisplatin; Drug: Placebo
- Phase 3 - Arm A or B (Experimental): Randomized 1:1 fianlimab (chosen dose) + cemiplimab + platinum-doublet chemotherapy
  Interventions: Drug: fianlimab; Drug: cemiplimab; Drug: Pemetrexed; Drug: Paclitaxel; Drug: Carboplatin; Drug: Cisplatin
- Phase 3 - Arm C (Experimental): Randomized 1:1 cemiplimab + platinum-doublet chemotherapy + placebo
  Interventions: Drug: cemiplimab; Drug: Pemetrexed; Drug: Paclitaxel; Drug: Carboplatin; Drug: Cisplatin; Drug: Placebo

INTERVENTIONS:
Drug: fianlimab — Administered intravenously (IV) every 3 weeks (Q3W)
  Other Names: REGN3767
  Arms: Phase 2 - Arm A; Phase 2 - Arm B; Phase 3 - Arm A or B
Drug: cemiplimab — Administered IV Q3W
  Other Names: REGN2810; Libtayo
Drug: Pemetrexed — IV Infusion, Q3W
  Other Names: Alimta
Drug: Paclitaxel — IV Infusion, Q3W
Drug: Carboplatin — IV Infusion, Q3W
  Other Names: Paraplatin
Drug: Cisplatin — IV infusion, Q3W
  Other Names: Platinol
Drug: Placebo — IV infusion, Q3W
  Arms: Phase 2 - Arm C; Phase 3 - Arm C

SUMMARY:
This study is researching an investigational drug called fianlimab (also called REGN3767) with two other medications called cemiplimab and chemotherapy, individually called a "study drug" or collectively called "study drugs". 'Investigational' means that the study drug is not approved for use outside of this study by any Health Authority. Examples of chemotherapy drugs include the following: Paclitaxel plus carboplatin, and Pemetrexed plus cisplatin. The study is being conducted in patients who have advanced non-small cell lung cancer (NSCLC).

The aim of the study is to see how effective the combination of fianlimab, cemiplimab, and chemotherapy is for treating advanced NSCLC, in comparison with cemiplimab and chemotherapy.

The study is looking at several other research questions, including:

* What side effects may happen from taking the study drugs
* How much of each study drug is in your blood at different times
* Whether the body makes antibodies against the study drugs (which could make the drug less effective or could lead to side effects)
* How administering the study drugs might improve your quality of life

ELIGIBILITY:
Key Inclusion Criteria:

1. Patients with non-squamous or squamous histology NSCLC with stage IIIB or stage IIIC disease who are not candidates for surgical resection or definitive chemoradiation per investigator assessment or stage IV (metastatic disease), who received no prior systemic treatment for recurrent or metastatic NSCLC.
2. Availability of an archival or on-study formalin-fixed, paraffin-embedded (FFPE) tumor tissue sample, without intervening therapy between biopsy collection and screening as described in the protocol
3. For enrollment in phase 2, patients should have PD-L1, expression results (regardless of expression level) determined by a College of American Pathologists (CAP)/Clinical Laboratory Improvement Amendments (CLIA) (or equivalently licensed, according to local regulations) accredited laboratory, as described in the protocol. For enrollment in phase 3, patients should have a valid PD-L1 result, regardless of expression level, using an assay as performed by a central laboratory, as described in the protocol.
4. At least 1 radiographically measurable lesion by computed tomography (CT) or magnetic resonance imaging (MRI) per RECIST 1.1 criteria. Target lesions may be located in a previously irradiated field if there is documented (radiographic) disease progression in that site.
5. Eastern Cooperative Oncology Group (ECOG) performance status of ≤1.
6. Adequate organ and bone marrow function as defined in the protocol.

Key Exclusion Criteria:

1. Active or untreated brain metastases or spinal cord compression. Patients are eligible if central nervous system (CNS) metastases are adequately treated and patients have neurologically returned to baseline (except for residual signs or symptoms related to the CNS treatment) for at least 2 weeks prior to enrollment. Patients must be off (immunosuppressive doses of) corticosteroid therapy.
2. Patients with tumors tested positive for actionable epidermal growth factor receptor (EGFR) gene mutations, anaplastic lymphoma kinase (ALK) gene translocations, or ROS oncogene 1 (ROS1) fusions, as described in the protocol.
3. Encephalitis, meningitis, or uncontrolled seizures in the year prior to enrollment.
4. History of interstitial lung disease (eg, idiopathic pulmonary fibrosis or organizing pneumonia), of active, noninfectious pneumonitis that required immune-suppressive doses of glucocorticoids to assist with management, or of pneumonitis within the last 5 years. A history of radiation pneumonitis in the radiation field is permitted as long as pneumonitis resolved ≥6 months prior to enrollment.
5. Known primary immunodeficiencies, either cellular (eg, DiGeorge syndrome, T-cell-negative severe combined immunodeficiency [SCID]) or combined T- and B-cell immunodeficiencies (eg, T- and B-cell negative SCID, Wiskott Aldrich syndrome, ataxia telangiectasia, common variable immunodeficiency).
6. Ongoing or recent (within 2 years) evidence of significant autoimmune disease that required treatment with systemic immunosuppressive treatments, which may suggest risk of immune-mediated treatment-emergent adverse events (imTEAEs). Patients with uncontrolled type 1 diabetes mellitus or with uncontrolled adrenal insufficiency are excluded. The following are not exclusionary: vitiligo, childhood asthma that has resolved, residual hypothyroidism that required only hormone replacement, or psoriasis that does not require systemic treatment.
7. Patients with a condition requiring corticosteroid therapy (>10 mg prednisone/day or equivalent) within 14 days of randomization. Physiologic replacement doses are allowed even if they are >10 mg of prednisone/day or equivalent, as long as they are not being administered for immunosuppressive intent. Patients with clinically relevant systemic immune suppression within the last 3 months before trial enrollment are excluded. Inhaled or topical steroids are permitted, provided that they are not for treatment of an autoimmune disorder.
8. Patients who have received prior systemic therapies are excluded with the exception of the following:

   1. Adjuvant or neoadjuvant platinum-based doublet chemotherapy (after surgery and/or radiation therapy) if recurrent or metastatic disease develops more than 6 months after completing therapy as long as toxicities have resolved to CTCAE grade ≤1 or baseline with the exception of alopecia and peripheral neuropathy.
   2. Anti-PD-(L)1 with or without LAG-3 as an adjuvant or neoadjuvant therapy as long as the last dose is >12 months prior to enrollment.
   3. Prior exposure to other immunomodulatory or vaccine as an adjuvant or neoadjuvant therapy such as Cytotoxic T-lymphocyte-associated protein 4 (anti-CTLA-4) antibodies as long as the last dose is >6 months prior to enrollment. Immune-mediated AEs must be resolved to CTCAE grade ≤1 or baseline by the time of enrollment. Endocrine immune-mediated AEs controlled with hormonal or other non-immunosuppressive therapies without resolution prior to enrollment are allowed.

Note: Other protocol-defined Inclusion/ Exclusion Criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 950 (Estimated)
Dates: Start 2023-08-08 (Actual); Primary Completion 2030-01-16 (Estimated); Study Completion 2031-12-23 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) as assessed by blinded independent review committee (BICR) using RECIST 1.1 | Up to 136 Weeks
  Phase 2 ORR is defined as proportion of patients with a best overall response of confirmed complete response (CR) or partial response (PR).
Overall Survival (OS) | Up to 5 years
  Phase 3 Defined as the time from randomization to the date of death due to any cause

SECONDARY OUTCOMES:
Incidence of treatment-emergent adverse event (TEAEs) | Up to 108 weeks
  Phase 2 & Phase 3 A TEAE is any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product, which does not necessarily have a causal relationship with this treatment
Incidence of treatment-related TEAEs | Up to 108 weeks
  Phase 2 & Phase 3
Incidence of serious adverse events (SAEs) | Up to 108 weeks
  Phase 2 & Phase 3
  Any untoward medical occurrence that at any dose:
  * Results in death - includes all deaths, even those that appear to be completely unrelated to study drug (eg, a car accident in which a patient is a passenger)
  * Is life-threatening
  * Requires in-patient hospitalization or prolongation of existing hospitalization • Results in persistent or significant disability/incapacity
  * Is a congenital anomaly/birth defect
  * Is an important medical event
Incidence of adverse events of special interest (AESIs) | Up to 108 weeks
  Phase 2 & Phase 3 Serious or non-serious; is one of scientific and medical concern specific to the sponsor's product or program, for which ongoing monitoring and rapid communication by the Investigator to the sponsor can be appropriate. Such an event might warrant further investigation in order to characterize and understand it.
Incidence of immune-mediated adverse events (imAEs) | Up to 108 weeks
  Phase 2 & Phase 3 Immune-mediated AEs are thought to be caused by unrestrained cellular immune responses directed at normal host tissues. An imAE can occur shortly after the first dose or several months after the last dose of treatment. Early detection and management reduces the risk of severe drug induced toxicity
Occurrence of interruption of study drug(s) due to AEs | Up to 108 weeks
  Phase 2 & Phase 3
Occurrence of discontinuation of study drug(s) due to AEs | Up to 108 weeks
  Phase 2 & Phase 3
Incidence of deaths due to TEAE | Up to 108 weeks
  Phase 2 & Phase 3
Incidence of grade 3-4 laboratory abnormalities | Up to 108 weeks
  Phase 2 & Phase 3
  ≥ grade 3 per National Cancer Institute-Common Terminology Criteria for Adverse Events [NCI-CTCAE v5.0]
ORR by investigator assessment using RECIST 1.1 | Up to 136 Weeks
  Phase 2 & Phase 3
Disease control rate (DCR) by BICR | Up to 136 Weeks
  Phase 2 and Phase 3 DCR is defined as CR + PR + stable disease (SD)
DCR by investigator assessment | Up to 136 Weeks
  Phase 2 and Phase 3 DCR is defined as CR + PR + stable disease (SD)
Time to tumor response (TTR) by BICR | Up to 136 Weeks
  Phase 2 and Phase 3 TTR is defined as the time from randomization to the date of the first response of CR or PR (whichever is first recorded) for patients with confirmed CR or PR.
TTR by investigator assessment | Up to 136 Weeks
  Phase 2 and Phase 3 TTR is defined as the time from randomization to the date of the first response of CR or PR (whichever is first recorded) for patients with confirmed CR or PR
Duration of response (DOR) by BICR | Up to 5 Years
  Phase 2 and Phase 3 DOR is defined as the time from first response of CR or PR to first radiographic progression or death due to any cause for patients with confirmed CR or PR
DOR by investigator assessment | Up to 5 Years
  Phase 2 and Phase 3 DOR is defined as the time from first response of CR or PR to first radiographic progression or death due to any cause for patients with confirmed CR or PR
Progression free survival (PFS) by BICR | Up to 5 Years
  Phase 2 and Phase 3 PFS is defined as the time from randomization to the date of the first radiographic progression or death due to any cause, whichever occurred earlier
PFS by investigator assessment | Up to 5 Years
  Phase 2 and Phase 3 PFS is defined as the time from randomization to the date of the first radiographic progression or death due to any cause, whichever occurred earlier
OS | Up to 5 Years
  Phase 2 Defined as the time from randomization to the date of death due to any cause
Change from baseline in patient-reported global health status/quality of life (GHS/QoL) per European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) | Up to 108 weeks
  Phase 2 & Phase 3 EORTC-QLQ-C30 is a 30-item subject self-report questionnaire composed of both multi-item and single scales, including a GHS/QoL scale. Participants rate items on a four-point scale, with 1 as "not at all" and 4 as "very much." A change of 5 - 10 points is considered a small change. A change of 10 - 20 points is considered a moderate change.
Change from baseline in physical functioning per EORTC QLQ-C30 | Up to 108 weeks
  Phase 2 & Phase 3
Change from baseline in patient-reported chest pain per European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Lung Cancer 13 (EORTC QLQ-LC13) | Up to 108 weeks
  Phase 2 & Phase 3 EORTC QLQ-LC 13 is a lung cancer specific module developed to assess lung cancer-associated symptoms and treatment-related side effects among lung cancer patients
Change from baseline in patient-reported dyspnea per EORTC QLQ-LC13 | Up to 108 weeks
  Phase 2 & Phase 3
Change from baseline in patient-reported cough per EORTC QLQ-LC13 | Up to 108 weeks
  Phase 2 & Phase 3
Time until definitive deterioration in patient-reported global health status/QoL per EORTC QLQ-C30 | Up to 108 weeks
  Phase 2 & Phase 3
Time until definitive deterioration in patient-reported physical functioning per EORTC QLQ-C30 | Up to 108 weeks
  Phase 2 & Phase 3
Time until definitive deterioration in patient-reported chest pain per EORTC QLQ-LC13 | Up to 108 weeks
  Phase 2 & Phase 3
Time until definitive deterioration in patient-reported dyspnea per EORTC QLQ-LC13 | Up to 108 weeks
  Phase 2 & Phase 3
Time until definitive deterioration in patient-reported cough per EORTC QLQ-LC13 | Up to 108 weeks
  Phase 2 & Phase 3
Time until definitive deterioration in a composite of these three symptoms: patient-reported chest pain, dyspnea and cough per EORTC QLQ-LC13 | Up to 108 weeks
  Phase 2 & Phase 3
Change from baseline in patient-reported general health status per EuroQoL 5-Dimensional 5-Level Scale (EQ-5D-5L) VAS | Up to 108 weeks
  Phase 2 & Phase 3 The EQ-5D-5L VAS records the respondent's self-rated health on a 10 centimeter (cm) vertical, visual analogue scale. It is rated by the respondent on a scale 0 to 100, with 0 being "the worst health you can imagine" and 100 being "the best health you can imagine".
Change from baseline in patient-reported severity with usual or daily activities due to fatigue per the Patient Reported Outcomes for Common Terminology Criteria for Adverse Events (PRO-CTCAE) | Up to 108 weeks
  Phase 2 & Phase 3 PRO-CTCAE questionnaire assesses side effect symptoms in cancer clinical trials using a PRO-CTCAE score. The PRO-CTCAE includes an item library of 124 items representing 78 symptomatic toxicities drawn from the CTCAE.
Change from baseline in patient-reported interference with usual or daily activities due to fatigue per the PRO-CTCAE | Up to 108 weeks
  Phase 2 & Phase 3
Concentrations of cemiplimab in serum | Up to 136 weeks
  Phase 2 & Phase 3
Concentrations of fianlimab in serum | Up to 136 weeks
  Phase 2 & Phase 3
Immunogenicity, as measured by anti-drug antibodies (ADA) to fianlimab | Up to 136 weeks
  Phase 2 & Phase 3
Immunogenicity, as measured by ADA to cemiplimab | Up to 136 weeks
  Phase 2 & Phase 3
Immunogenicity, as measured by neutralizing antibodies (NAb) to fianlimab | Up to 136 weeks
  Phase 2 & Phase 3
Immunogenicity, as measured by NAb to cemiplimab | Up to 136 weeks
  Phase 2 & Phase 3

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (76):
- United States (29):
  - Arizona Clinical Research Center, Tucson, Arizona
  - Yuma Regional Medical Center, Yuma, Arizona
  - The Oncology Institute of Hope & Innovation, Cerritos, California
  - Crosson Cancer Institute, Fullerton, California
  - St. Joseph Hospital Orange, Orange, California
  - Desert Hematology Oncology Medical Group Incorporated, Rancho Mirage, California
  - Emad Ibrahim, MD, Inc., Redlands, California
  - PIH Health Hospital, Whittier, California
  - Rocky Mountain Regional VA Medical Center, Aurora, Colorado
  - Yale Cancer Center, New Haven, Connecticut
  - Clermont Oncology Center, Clermont, Florida
  - Miami Veterans Administration HealthCare System, Miami, Florida
  - Mid Florida Hematology and Oncology Center, Orange City, Florida
  - Tallahassee Memorial Healthcare, Tallahassee, Florida
  - University of Illinois, Chicago, Illinois
  - Northwest Oncology and Hematology, Rolling Meadows, Illinois
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - Hattiesburg Clinic, Hattiesburg, Mississippi
  - Capital Health Hopewell Medical Center, Pennington, New Jersey
  - New Mexico Cancer Care Alliance, Albuquerque, New Mexico
  - NYU Langone Health Perlmutter Cancer Center, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Clinical Research Alliance Inc, Westbury, New York
  - Gabrail Cancer Center Research, Canton, Ohio
  - Thompson Cancer Survival Center (TCSC ) - Downtown, Knoxville, Tennessee
  - University of Tennessee Medical Center, Knoxville, Tennessee
  - University of Virginia Medical Center, Charlottesville, Virginia
  - Bon Secours Cancer Institute Richmond, Midlothian, Virginia
- Australia (6):
  - Macquarie University Health Science Center (MQ Health), Macquarie Park, New South Wales
  - Southern Medical Day Care Centre, Wollongong, New South Wales
  - Ballarat Regional Integrated Cancer Centre (BRICC), Ballarat, Victoria
  - Bendigo Hospital, Bendigo, Victoria
  - St Vincents Hospital Melbourne, Fitzroy, Victoria
  - St John of God Murdoch Hospital, Murdoch, Western Australia
- Canada (2):
  - British Columbia Cancer Center-Kelowna, Kelowna, British Columbia
  - Hopital Cite de la Sante, Laval, Quebec
- Georgia (10):
  - LLC High-Tech Hospital Medcenter, Batumi, Adjara
  - Israeli Georgian Medical Research Clinic Helsicore, Tbilisi
  - Research Institute of Clinical Medicine, Tbilisi
  - LTD New Hospitals, Tbilisi
  - High Technology Medical Center, University Clinic Tbilisi, Tbilisi
  - LTD Archangel St. Michael Multiprofile Clinical Hospital, Tbilisi
  - NNLE New Vision University Hospital, Tbilisi
  - The Institute of Clinical Oncology, Tbilisi
  - TIM - Tbilisi Institute of Medicine, Tbilisi
  - JSC Evex Hospitals - Caraps Medline, Tbilisi
- Israel (2):
  - Sheba Medical Center, Ramat Gan, Central District
  - Assuta Medical Centers, Tel Aviv
- Malaysia (7):
  - Hospital Sultan Ismail, Johor Bahru, Johor
  - Hospital Kuala Lumpur, Kuala Lumpur, Kuala Lumpur
  - Hospital Tengku Ampuan Afzan (HTTA), Kuantan, Pahang
  - Mount Miriam Cancer Hospital, Tanjung Bungah, Pulau Pinang
  - National Cancer Institute, Putrajaya, Putrajaya
  - Sarawak General Hospital, Kuching, Sarawak
  - Hospital Pulau Pinang, Pulau Pinang
- South Korea (10):
  - CHA Bundang Medical Center CHA University, Seongnam-si, Gyeonggi-do
  - St. Vincents Hospital - The Catholic University of Korea, Suwon, Gyeonggi-do
  - Ajou University Hospital, Suwon, Gyeonggi-do
  - Gachon University Gil Medical Center, Incheon, Namdong-gu
  - Chungbuk National University Hospital, Cheongju-si, North Chungcheong
  - Chungnam National University Hospital, Daejeon
  - Inha University Hospital, Incheon
  - Asan Medical Center, Seoul
  - Korea University Guro Hospital, Seoul
  - Ulsan University Hospital, Ulsan
- Taiwan (8):
  - Dalin Tzu Chi Hospital, Dalin Town, Chiayi
  - Buddhist Tzu Chi General Hospital, Hualien City, Hualien
  - Chung-Ho Memorial Hospital, Kaohsiung City
  - Taipei Medical University - Shuang Ho Hospital, New Taipei City
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Taipei Medical University Hospital, Taipei
  - Tri-Service General Hospital, Taipei
- Lampang Cancer Center, Lampang, Changwat Lampang, Thailand
- Adana City Education and Research Hospital, Adana, Yuregir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
All Individual Patient Data (IPD) that underlie publicly available results will be considered for sharing
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: When Regeneron has:
  * received marketing authorization from major health authorities (e.g., FDA, European Medicines Agency (EMA), Pharmaceuticals and Medical Devices Agency (PMDA), etc.) for the product and indication or has globally discontinued development of the product for all indications on or after April 2020 and has no plans for future development
  * made the study results publicly available (e.g., scientific publication, scientific conference, clinical trial registry)
  * the legal authority to share the data, and
  * ensured the ability to protect participant privacy.
Access Criteria: Qualified researchers can submit a proposal for access to individual patient or aggregate level data from a Regeneron-sponsored clinical trial through Vivli. Regeneron's Independent Research Request Evaluation Criteria can be found at: https://www.regeneron.com/sites/default/files/Regeneron-External-Data-Sharing-Policy-and-Independent-Research-Request-Evaluation-Criteria.pdf
URL: https://vivli.org/